CLINICAL TRIAL: NCT07336316
Title: Multimodal Cardiovascular Magnetic Resonance Imaging for Cardiometabolic Pre-HF and HFpEF: Integrated Phenotyping, Precision Diagnosis, and Risk Stratification
Brief Title: Multimodal Cardiovascular Magnetic Resonance Imaging for Cardiometabolic Pre-HF and HFpEF
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-CMHF
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes (DM); Hypertension; Heart Failure; Obesity & Overweight
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Heart Failure; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study aiming to characterize the pathophysiological features and clinical significance of cardiometabolic early-stage heart failure using advanced multimodal cardiovascular magnetic resonance (CMR) imaging. The study will focus on patients with cardiometabolic risk factors such as diabetes, hypertension, and obesity who are in the pre-heart failure (pre-HF) stage or have heart failure with preserved ejection fraction (HFpEF). The study seeks to establish a full-chain imaging framework-from precise phenotypic classification and sensitive noninvasive diagnosis to individualized cardiovascular risk stratification. Participants will undergo multimodal CMR scans and comprehensive clinical evaluations and be followed up for primary outcome.

DETAILED DESCRIPTION:
Advanced noninvasive multimodal cardiovascular magnetic resonance (CMR) imaging techniques-including early functional impairment detection (feature tracking), myocardial tissue characterization (T1 mapping), hemodynamic changes (hemodynamic force [HDF] analysis), and magnetic resonance spectroscopy-have significant potential clinical value, especially for capturing the complex pathophysiology of cardiometabolic early-stage heart failure.

This study applies these advanced CMR imaging techniques to individuals with cardiometabolic risk factors and early-stage heart failure (pre-HF and HFpEF) to perform multidimensional, comprehensive CMR analyses. The goal is to identify characteristic imaging patterns for this cohort, develop targeted diagnostic models, facilitate their application in risk prediction and individualized management, and ultimately establish an imaging evaluation framework that can optimize clinical pathways for cardiometabolic pre-HF and HFpEF.

This study enrolls patients undergoing CMR who have early-stage cardiometabolic heart failure (pre-HF and HFpEF), including with diabetes, hypertension, obesity and so on. Clinical data, laboratory results, and echocardiographic parameters will be collected.

Through cross-sectional analysis, the study will evaluate chamber structure and function, myocardial tissue characteristics, hemodynamics, and myocardial energy metabolism, and summarize characteristic imaging phenotypes of cardiometabolic early-stage heart failure. Imaging parameters will be compared to identify robust noninvasive diagnostic markers and optimize the diagnostic framework for cardiometabolic early-stage heart failure. In addition, participants will be followed longitudinally to collect outcome events. The predictive value of CMR-derived indicators for clinical outcomes will be analyzed, and risk prediction models will be developed to achieve precise risk stratification for patients with early-stage cardiometabolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≥ 50%；
* Presence of cardiovascular risk factors, including, but not limited to, the following: diabetes mellitus, hypertension, obesity.

Exclusion Criteria:

* Primary cardiomyopathy (e.g., hypertrophic, dilated, and restrictive cardiomyopathy)
* Acute coronary syndrome in the previous 30 days
* More than moderate valvular disease
* Restrictive pericardial disease
* Severe arrhythmia
* Heart tumors
* Infiltrative cardiomyopathy (e.g., cardiac amyloidosis)
* Congenital heart disease
* Poor image quality insufficient for delineating the endocardium and epicardium

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: early-stage heart faliure with cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of all cause or cardiovascular death | 2-15 years
Incidence Rate of HF hospitalization | 2-15 years
  HF hospitalization was defined as an unplanned hospitalization with documented clinical and radiological evidence for HF and need for diuretic treatment

OTHER OUTCOMES:
Incidence Rate of newly onset heart failure | 2-15 years

REFERENCES:
- [Result] McHugh K, DeVore AD, Wu J, Matsouaka RA, Fonarow GC, Heidenreich PA, Yancy CW, Green JB, Altman N, Hernandez AF. Heart Failure With Preserved Ejection Fraction and Diabetes: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Feb 12;73(5):602-611. doi: 10.1016/j.jacc.2018.11.033. PMID 30732715
- [Result] Smiseth OA, Morris DA, Cardim N, Cikes M, Delgado V, Donal E, Flachskampf FA, Galderisi M, Gerber BL, Gimelli A, Klein AL, Knuuti J, Lancellotti P, Mascherbauer J, Milicic D, Seferovic P, Solomon S, Edvardsen T, Popescu BA; Reviewers: This document was reviewed by members of the 2018-2020 EACVI Scientific Documents Committee. Multimodality imaging in patients with heart failure and preserved ejection fraction: an expert consensus document of the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2022 Jan 24;23(2):e34-e61. doi: 10.1093/ehjci/jeab154. PMID 34729586
- [Result] Obokata M, Reddy YNV, Pislaru SV, Melenovsky V, Borlaug BA. Evidence Supporting the Existence of a Distinct Obese Phenotype of Heart Failure With Preserved Ejection Fraction. Circulation. 2017 Jul 4;136(1):6-19. doi: 10.1161/CIRCULATIONAHA.116.026807. Epub 2017 Apr 5. PMID 28381470
- [Result] Daou D, Tong D, Schiattarella GG, Gillette TG, Hill JA. What Is Cardiometabolic HFpEF and How Can We Study it Preclinically? JACC Basic Transl Sci. 2025 Oct;10(10):101295. doi: 10.1016/j.jacbts.2025.04.009. Epub 2025 Jul 30. PMID 40742364